CLINICAL TRIAL: NCT06621264
Title: EXercise ACTivity to Improve Mobility, Active Behavior and Quality of Life of Chronic Kidney Disease Patients With Peripheral Artery Disease: the EXACTckd-pad Multicenter Randomized Controlled Trial
Brief Title: Exercise Activity to Improve Mobility in Patients With CKD and PAD
Acronym: EXACT-CKDPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: University of Verona, Italy (Unknown); Reggio Calabria (Other)
Responsible Party: Principal Investigator, Fabio Manfredini, Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNRR-MAD-2022-12376611
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease Stage 3 and 4; Peripheral Artery Disease (PAD)
Keywords: Exercise therapy;; Mobility; Ageing; Chronic Kidney Disease; Peripheral artery disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Peripheral Arterial Disease | interventions — Exercise; Dosage Forms; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Patients enrolled in this group will receive a detailed 6-month exercise prescription aimed at providing in-home low fatiguingwalking training (at light-moderate intensity, or 2-3 out of 10 of the CR10 Borg's scale). The program consists of a two daily 10-minute interval walking sessions (1 minute walking : 1 minute resting) at a prescribed speed controlled by a digital metronome (https://www.youtube.com/watch?v=ki8YX_t-0jA). The training speed will be set up according to the patients baseline walking capacity (approximately 50% lower than the habitual gait speed) and will be weekly increased until reaching the habitual gait speed. The training time will be maintained constant throughout the entire program.
  Exercise prescription will be updated during two intermediate hospital visits at the 1st and 3rd months. Patients will be provided with a digital application properly developed to keep pacing and to record the correct training execution.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Control group (Placebo Comparator): Patients enrolled in the Co group will receive standard CKD-PAD care, including optimal medical therapy and nutritional advices
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Patients enrolled in this group will receive a detailed 6-month exercise prescription aimed at providing in-home low fatiguing walking training (at light-moderate intensity, or 2-3 out of 10 of the CR10 Borg's scale). The program consists of a two daily 10-minute interval walking sessions (1 minute walking : 1 minute resting) at a prescribed speed controlled by a digital metronome (https://www.youtube.com/watch?v=ki8YX_t-0jA). The training speed will be set up according to the patients baseline walking capacity (approximately 50% lower than the habitual gait speed) and will be weekly increased until reaching the habitual gait speed. The training time will be maintained constant throughout the entire program. Exercise prescription will be updated during two intermediate hospital visits at the 1st and 3rd months. Patients will be provided with a digital application properly developed to keep pacing and to record the correct training execution.
  Other Names: exercise; rehabilitation
  Arms: Exercise group
Other: Control (Standard treatment) — Patients enrolled in the Co group will receive standard CKD-PAD care, including optimal medical therapy and nutritional advices
  Other Names: Usual care
  Arms: Control group

SUMMARY:
People affected by chronic kidney disease and concomitant diagnosed peripheral artery disease at intermediate stages, without contraindications to exercise therapy will be invited to participate in the study.

Whose providing informed consent, will be randomly assigned to one of two groups:

1. Exercise program receiving two daily 10-minute interval walking sessions at a slow increasing speed.
2. Control group: receiving usual care including optimal medical therapy and nutritional advice.

Patients of both groups will be measured at baseline, after the end of the exercise program (6-month) and at follow up (12-month). Outcome measures will include walking ability by the 6-minute walking test (primary outcome) and lower limbs perfusion, body composition, quality of life, laboratory outcomes and long-term hospitalizations.

DETAILED DESCRIPTION:
People with chronic kidney disease (CKD) are exposed to a high risk of developing peripheral artery disease (PAD) and its related adverse health outcomes. This dangerous combination of pathological conditions increases overall cardiovascular risk, mortality and lower limbs amputations.

The scientific literature suggests a strategic co-management of CKD-PAD patients by multidisciplinary teams including specialists of different areas and expertise. Indeed, a common issue is that both these diseases are negatively associated with a sedentary behavior. Exercise therapy may enhance the physical functioning, the risk factors management, the lower limbs vascularization and reduce the cardiovascular risk that affects this population. Since the CKD-PAD population is less likely to be provided recommended optimal care, and considering that 2 out of 3 CKD patients have a completely sedentary behavior for several barriers to training participation, proper exercise programs should be developed. This multicenter randomized-controlled trial aims to test the effectiveness of a 6-month home-based structured walking program on physical functioning and laboratory and clinical outcomes. Purposely 100 CKD patients at KDOQI stages III or IV with concomitant PAD at Rutherford's stages I to III, aged > 18 years and without absolute contraindications to exercise training will be randomized to receive an exercise intervention (Ex) or usual care (Control, Co). The 6-month training intervention, previously tested in PAD and CKD patients, consist in two 10-minute daily interval walking sessions performed inside the home.

Patients will receive a detailed exercise prescription according to their baseline walking capacity, with the walking speed maintained at home through sound pacing by a digital metronome. The prescribed speed will be weekly increased from the 60 to the 100% of their baseline walking speed with a fixed working time throughout the program. Two serial visits during the program will be scheduled to reinforce adherence to exercise, maintained and verified by a digital application, and to control the blood pressure. Patients enrolled in the Co group will receive standard CKD-PAD care, including optimal medical therapy and nutritional advices.

The primary outcome of the study will be the variations of mobility as assessed by the 6-minute walking test at the end of the program. Secondary outcomes will include lower limbs perfusion and strength, body composition and bone mineral density, quality of life, laboratory outcomes including rate of progression of CKD and the long-term hospitalizations and mortality.

Outcome measures will be assessed by blinded operators at baseline, at the end of the program for exercise group (6-month) and at 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease at KDOQI stages III or IV and concomitant Peripheral artery disease at stages I, II, III;
* ability to walk independently;
* cognitive function to give informed consent identified by a Mini Mental Status Examination score greater or equal to 20/30
* absence of clinical conditions contraindicating exercise therapy (e.g., unstable angina, severe heart failure at NYHA class IV, anemia with lower than 10.0 g/dl).

Exclusion Criteria:

* major amputations;
* major surgery planned in the next 3 months;
* known comorbid conditions that may limit survival to less than 2 years;
* inability or unwillingness to comply with protocol requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walking test | Baseline; End of program (6-month); Follow up (12-month)
  The patients will be instructed to walk back and forth on a 20-meter corridor aiming at covering as much distance as possible. The total distance covered (6MWD) will be measured in meters

SECONDARY OUTCOMES:
Lower limbs perfusion | Baseline; end of the program (6-month); Follow up (12-month).
  This measure will be performed according to the published standards with the patient laying by dividing the blood pressure at the ankle with the systolic blood pressure.
handgrip strength will be measured by a standard dynamometer | Baseline; end of the program (6-month); Follow up (12-month).
  both hands, patients will be asked to perform three repetitions. The peak and mean values are collected
Quality of life will be assessed by the short-form 36 (SF-36) questionnaire | Baseline; end of the program (6-month); Follow up (12-month).
  This is a generic questionnaire that contains 36 questions referring to 8 specific domains related to patient health over the previous 4 weeks
Bone mineral density | Baseline; end of the program (6-month); Follow up (12-month).
  bone mineral density will be measured through phalangeal quantitative ultrasound with an ultrasound signal of 1.25 MHz frequency and a methodology devoid of X-rays. The results are consistent with those obtained by standard DEXA
lower limbs strength assessed by the 5-time sit-to-stand test | Baseline; end of the program (6-month); Follow up (12-month).
  Patients will raise up from a standard height chair with their arms folded across the chest five times as quickly as possible. The total time elapsed for completing the five repetitions is recorded in seconds
Body mass index | Baseline, end of the program (6-month); follow up (12-month)
  Body composition will be assessed with direct measures of height and weight. Body mass index will be calculated as the ratio between weight (in kg) and the squared height (in meters)
Circulating indexes of kidney function | Baseline, end of treatment (6-month); follow up (12-month)
  Serum creatinine will be directly measured through standard laboratory methods. The estimated glomerular filtration rate will be calculated through the 2009 Chronic Kidney Disease Epidemiology Collaboration equation
Long-term survival rate | Baseline, end of treatment (6-month); follow up (12-month); follow up (18-month); Follow up (24-month); FOllow up (36-month)
  All-cause mortality of the enrolled patients will be checked from the regionals datasets. In case of positive findings, the days elapsed from enrollment to the event will be recorded for additional analyses, as well as the reasons and the diagnoses.
Long-term hospitalizations | Baseline, end of treatment (6-month); follow up (12-month); follow up (18-month); Follow up (24-month); FOllow up (36-month)
  All-cause hospitalization will be checked from the regionals datasets. In case of positive findings, the days elapsed from enrollment to the event will be recorded for additional analyses, as well as the reasons and the diagnoses.
Rate of admission to dialysis | Baseline, end of treatment (6-month); follow up (12-month); follow up (18-month); Follow up (24-month); FOllow up (36-month)
  Number of patients that will be admitted to dialysis will be recorded and the time from enrollment to the dialysis admission will calculated
Pain-free walking distance | Baseline, end of treatment (6-month), follow up (12-month)
  During the 6-minute walking test, the distance at the onset of symptoms referred by the patient will be collected and reported

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Manfredini Prof. Roberto Manfredini, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (3):
- Italy (3):
  - University Hospital of Ferrara, Ferrara, Italy
  - Ospedale Pederzoli Peschiera del Garda, Peschiera del Garda, Italy
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria, Italy

IPD SHARING:
Plan to Share IPD: Yes
The database generated for the study with anonimyzed patients' characteristics will be available on institution public repository
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol, along with the statistical analysis plan will be available when published on an open access journal.

REFERENCES:
- [Derived] Manfredini F, Panuccio V, Battaglia Y, Storari A, Lamberti N, Piva G, Veronesi M, Tripepi R, Rinaldo N, Crepaldi A, Momente C, Piccinini A, Traina L, Fargion AT, Straudi S, Baroni A, De Giorgi A, Martinuzzi C, Monesi M, Capitanini A, Aucella F, Cupisti A, Mallamaci F, Zoccali C, Manfredini R. Exercise therapy to improve mobility, active behaviour and quality of life of chronic kidney disease patients with peripheral artery disease: study protocol for the EXACT-CKDPAD multicentre randomised controlled trial. BMJ Open Sport Exerc Med. 2025 Jul 15;11(3):e002740. doi: 10.1136/bmjsem-2025-002740. eCollection 2025. PMID 40672525